CLINICAL TRIAL: NCT05081037
Title: Lifestyle Interventions to Prevent Postpartum Type II Diabetes Mellitus in Asian Women With a History of Gestational Diabetes Mellitus
Brief Title: Integrated Hyperglycaemia Incentivised Postnatal Surveillance Study (I-HIPS)
Acronym: I-HIPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Duke-NUS Graduate Medical School (Other); Institute for Human Development and Potential (IHDP), Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020/3070
Record Dates: First submitted 2021-09-23; First posted 2021-10-18 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Gestational Diabetes; Glucose Metabolism Disorders; Metabolic Disease
Keywords: gestational diabetes; post-partum intervention; Body composition
MeSH Terms: conditions — Diabetes, Gestational; Glucose Metabolism Disorders; Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: Participants randomized to both the control (Scheduled Care Group) and the intervention group (Wearable Care Group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wearable Care Group (Experimental): This group will receive both a continous glucose monitoring sensor and an exercise tracker to be worn for at least 2 weeks at each study visit timepoint.
  Interventions: Device: Wearable Care Group
- Scheduled Care Group (No Intervention): This group will receive standard medical care with dietary and nutritional advice alone.

INTERVENTIONS:
Device: Wearable Care Group — Continous glucose monitoring sensor: Study participants wear the sensor on the back of either right or left upper arm for up to 14 days. Glucose levels will be recorded from the interstitial fluid every 15 minutes using intermittent/ flash glucose scanning.
  Exercise tracker: A FitBit watch will be given to the participants for use to track physical activity levels.
  Arms: Wearable Care Group

SUMMARY:
This study aims to test the following hypotheses in a randomized controlled trial of post-partum women with a history of gestational diabetes mellitus (GDM) that will be followed up for up to 4 years:

1. Post-partum pregnancy is ideal for behavioural modification and adopting a healthy lifestyle. Using the continous glucose monitoring (CGM) sensor and an exercise tracker will promote self-motivation and awareness by positive reinforcement and behavioural changes to improve diet, control body weight and increase physical activity in this group of post-partum women who are at high risk for developing Type II Diabetes.
2. The use of the continous glycose monitoring (CGM) sensor and exercise tracker will motivate women to modify their dietary food intake and physical activity over time, reducing their cardiovascular risk factors for developing metabolic syndrome by lowering their baseline blood pressure, BMI, reducing their waist circumference and body fat mass, glycaemic levels and fasting lipids within the targeted healthy range.
3. There will be an increase in the quality adjusted life years (QALYs) gained based on improvements in HbA1C and other proximal outcomes at the end of the trial.

DETAILED DESCRIPTION:
The increased incidence of gestational diabetes mellitus (GDM) resulting from increased insulin resistance has become a major health concern. GDM affects 5-10% of pregnant women in Europe, while the prevalence in Asian populations is significantly higher at approximately 15-20%. There is a need for early postpartum intervention strategies beginning soon after birth, but yet there are limited of such intervention studies conducted in Asia.

This is a randomized controlled trial and hospital-based study. A total of 300 post-partum women who attended KK Women's and Children's Hospital (KKH) for antenatal consultation and were diagnosed with GDM using International association of diabetes and pregnancy study groups (IADPSG) guidelines at KKH, with a BMI range from 20-40, and physically fit to participate in moderate intensity walking will be approached for prospective recruitment. These subjects will be followed-up to determine if they will have normal oral glucose tolerance test (OGTT) results at 6 weeks postpartum. If all the inclusion criteria is met, these women will be recruited into the study.

The recruited women will be randomly allocated to the intervention or control group. Those placed in the intervention group, which will also be known as the Wearable Care Group, will receive both a continous glucose monitoring (CGM) and an exercise tracker which will be a FitBit watch. Those placed in the control group, which will also be known as the Scheduled Care Group will receive standard medical care.

Participants randomized to both the control (Scheduled Care Group) and the intervention group (Wearable Care Group) will be followed up in the specialist outpatient clinics with a total of 7 visits for up to 4 years. Various testing will be carried out at relevant time points.

Data will be collected through questionnaires and clinical measurements. The questionnaires include socio-economic factors, a quality of life questionnaire, maternal diet, medical histories, lifestyle factors, health status, and home environment. Bio-physical measurements will be obtained from anthropometric measurements of participants, human biological materials such as blood, are collected from the participants at their follow-up time points with the I-HIPS study upon their consent.

ELIGIBILITY:
Inclusion Criteria:

1. Women diagnosed antenatally with GDM by IADPSG criteria (15)
2. Normal 6 weeks post-natal OGTT
3. BMI range from 20-40
4. Physically fit to participate in moderate intensity walking

Exclusion Criteria:

1. Women with serious skin conditions (e.g. eczema) that precludes wearing the sensor for 14 days
2. Women who have any other serious chronic disease such as chronic kidney disease and heart disease

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2026-05-26 (Estimated); Study Completion 2026-05-26 (Estimated)

PRIMARY OUTCOMES:
Clinically diagnosed Type II Diabetes Mellitus | At 6 months (23-26 weeks) from baseline visit
  Clinical outcomes of Type II Diabetes Mellitus development determined by oral glucose tolerance test
Clinically diagnosed Type II Diabetes Mellitus | At 10-14 months from baseline visit
  Clinical outcomes of Type II Diabetes Mellitus development determined by oral glucose tolerance test
Clinically diagnosed Type II Diabetes Mellitus | At 22-26 months from baseline visit
  Clinical outcomes of Type II Diabetes Mellitus development determined by oral glucose tolerance test
Clinically diagnosed Type II Diabetes Mellitus | At 34-38 months from baseline visit
  Clinical outcomes of Type II Diabetes Mellitus development determined by oral glucose tolerance test
Body mass index at the end of the 6 month intervention period | At 6 months (23-26 weeks) from baseline
  Using weight and height measures
Body fat mass at the end of the 6 month intervention period | At 6 months (23-26 weeks) from baseline
  Measured using the bioelectrical impedance analysis scale

SECONDARY OUTCOMES:
Change in total energy intake from baseline at 6 months (23-26 weeks) | Baseline and 6 months (23-26 weeks)
  Assess the effect of continous glucose monitoring sensor use on total energy intake calculated using data captured from the 24-Hour recall food diary.
Change in total energy intake from baseline, 6 months, 12 months, 24 months and 36 months | Baseline, 6 months (23-26 weeks), 12 months (10-14 months), 24 months (22-26 months) and 36 months (34-38 months)
  Assess the effect of continous glucose monitoring sensor use on total energy intake captured using data captured from the 24-Hour recall food diary.
Change in diet quality from baseline at 6 months (23-26 weeks) | Baseline and 6 months (23-26 weeks)
  Assess the effect of continous glucose monitoring sensor use on diet quality derived using a 24-Hour recall food diary.
Change in diet quality from baseline, 6 months,12 months, 24 months and 36 months | Baseline, 6 months (23-26 weeks), 12 months (10-14 months), 24 months (22-26 months) and 36 months (34-38 months)
  Assess the effect of continous glucose monitoring sensor use on diet quality derived using a 24-Hour recall food diary.
Change in physical activity from baseline at 6 months (23-26 weeks) | Baseline and 6 months (23-26 weeks)
  Assess the effect of exercise tracker use on frequency and duration of physical activity using self-reported data from the International Physical Activity Questionnaire (IPAQ)
Change in physical activity from baseline, 6 months, 12 months, 24 months and 36 months | Baseline, 6 months (23-26 weeks), 12 months (10-14 months), 24 months (22-26 months) and 36 months (34-38 months)
  Assess the effect of exercise tracker use on frequency and duration of physical activity using self-reported data from the International Physical Activity Questionnaire (IPAQ)
Change in diastolic and systolic blood pressure measures from baseline at 6 months (23-26 weeks) | Baseline and 6 months (23-26 weeks)
  Using diastolic and systolic blood pressure measures
Change in diastolic and systolic blood pressure measures from baseline, 6 months, 12 months, 24 months and 36 months | Baseline, 6 months (23-26 weeks), 12 months (10-14 months), 24 months (22-26 months) and 36 months (34-38 months)
  Using diastolic and systolic blood pressure measures
Change in body mass index measures from baseline at 6 months (23-26 weeks) | Baseline and 6 months (23-26 weeks)
  Calculating body mass index using height and weight measures
Change in body mass index measures from baseline, 6 months, 12 months, 24 months and 36 months | Baseline, 6 months (23-26 weeks), 12 months (10-14 months), 24 months (22-26 months) and 36 months (34-38 months)
  Calculating body mass index using height and weight measures
Change in waist circumference measures from baseline at 6 months (23-26 weeks) | Baseline and 6 months (23-26 weeks)
  Using waist circumference measures
Change in waist circumference measures from from baseline, 6 months, 12 months, 24 months and 36 months | Baseline, 6 months (23-26 weeks), 12 months (10-14 months), 24 months (22-26 months) and 36 months (34-38 months)
  Using waist circumference measures
Change in body fat mass measures from baseline at 6 months (23-26 weeks) | Baseline and 6 months (23-26 weeks)
  Using body fat mass measured using the bioelectrical impedance analysis scale
Change in body fat mass measures from baseline, 6 months, 12 months, 24 months and 36 months | Baseline, 6 months (23-26 weeks), 12 months (10-14 months), 24 months (22-26 months) and 36 months (34-38 months)
  Using body fat mass measured using the bioelectrical impedance analysis scale
Change in HbA1c measures from baseline at 6 months (23-26 weeks) | Baseline and 6 months (23-26 weeks)
  Using HbA1c levels measured from blood samples
Change in HbA1c measures from baseline, 6 months, 12 months, 24 months and 36 months | Baseline, 6 months (23-26 weeks), 12 months (10-14 months), 24 months (22-26 months) and 36 months (34-38 months)
  Using HbA1c levels measured from blood samples
Change in fasting lipid profile from baseline at 6 months (23-26 weeks) | Baseline and 6 months (23-26 weeks)
  Using fasting lipid profiles (total cholesterol, Low-density lipoprotein (LDL) cholesterol, High-density lipoprotein (HDL) cholesterol, triglycerides) of blood samples
Change in fasting lipid profile from baseline, 6 months, 12 months, 24 months and 36 months | Baseline, 6 months (23-26 weeks), 12 months (10-14 months), 24 months (22-26 months) and 36 months (34-38 months)
  Using fasting lipid profiles (total cholesterol, Low-density lipoprotein (LDL) cholesterol, High-density lipoprotein (HDL) cholesterol, triglycerides) of blood samples

OTHER OUTCOMES:
Change in quality of life from baseline at 12 months (10-14 months) | Baseline and 12 months (10-14 months) and 36 months (34-38 months)
  Quality of life score measured using the EQ-5D-5L instrument
Change in quality of life from baseline at 36 months (34-38 months) | Baseline and 36 months (34-38 months)
  Quality of life score measured using the EQ-5D-5L instrument

CONTACTS AND LOCATIONS:
Overall Officials: Kok Hian Tan, MD, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No